CLINICAL TRIAL: NCT00219999
Title: Hepatitis C Virus and the Humoral Immune System
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LDU-0437; R01AI060561 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis; Hepacivirus; B Lymphocytes; Chemokines; Antibodies
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- HCV infection: current HCV infection, including intravenous drug users
- cryoglobulinemia: cryoglobulinemia and without HCV infection
- chronic liver disease: chronic liver disease not due to hepatitis C virus infection
- Sustained Virologic responders: successfully treated for HCV infection
- normal: normal, healthy volunteers

SUMMARY:
The purpose of this study is to measure specific chemokines, antibodies, and antibody-producing B cells in the blood of patients with hepatitis C virus (HCV) infection. Our hypothesis is that changes in chemokine levels affect the development of an effective immune response against HCV.

DETAILED DESCRIPTION:
The long-term goal of our research is to understand why immune complexes (ICs) are produced in patients infected with HCV, and whether these complexes affect virus interaction with target cells. We have found that many patients infected with HCV have an increased frequency of circulating B cells, but no evidence that the increased B cells are activated of proliferating. One possible mechanism for such an increase would be a change in levels of chemokines that influence B cell localization and trafficking. Our studies are aimed at testing the following hypotheses:

1. One hypothesis is that HCV infection results in increased levels of specific cytokines and chemokines that may affect the motility and localization of immature and mature B cells. An alternative model is that HCV infection leads to chronic antigenic stimulation of B lymphocytes, and that the abnormalities of B cell function associated with HCV infection reflect this chronic antigenic stimulation.
2. A second hypothesis is that autoantibodies and immune complexes present in HCV patient serum contribute to the persistence and spread of viral infection.

To test these hypotheses, we are measuring levels of chemokines, the frequency of circulating B cells (mature resting B cells, mature activated B cells, memory B cells, and immature B cells), and the levels and components of ICs in the blood of HCV-infected patients. Controls include healthy volunteers and patients with chronic liver disease unrelated to HCV infection. No interventions in patient care are planned. When patients elect to undergo standard antiviral therapies under the supervision of their hepatologists, we will study the outcomes of therapy (no virologic response, partial or transient virologic response, sustained virologic response) to determine whether any of the observed alterations in chemokine levels, B cell frequency or activation, or immune complex levels correlate with the patient's response to antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, no liver disease
* Chronic infection with hepatitis C virus
* Other chronic liver disease unrelated to hepatitis C virus
* Subjects in all groups must have sufficiently healthy veins to allow blood collection.

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigators, precludes the patient's participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinics of doctors at NYPH and the NYC metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2001-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Define the relationships between HCV infection, B cell phenotype, and B cell function | 5 years
  Define the relationships between HCV infection, B cell phenotype, and B cell function

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Dustin, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hosital, New York, New York, United States

REFERENCES:
- [Derived] Charles ED, Green RM, Marukian S, Talal AH, Lake-Bakaar GV, Jacobson IM, Rice CM, Dustin LB. Clonal expansion of immunoglobulin M+CD27+ B cells in HCV-associated mixed cryoglobulinemia. Blood. 2008 Feb 1;111(3):1344-56. doi: 10.1182/blood-2007-07-101717. Epub 2007 Oct 17. PMID 17942751
- See also: Related Info — http://www.rucares.org/clinicalstudies/list.php